CLINICAL TRIAL: NCT02068846
Title: BK Virus in Salivary Gland Disease
Brief Title: BK Virus in Salivary Gland Disease: Treating the Potential Etiologic Agent
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-0036; 1R21DE023046-01A1 (NIH)
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-06

CONDITIONS: HIV; Salivary Gland Disease; Benign Lymphoepithelial Lesion
Keywords: HIV; Salivary Gland Disease; Benign Lymphoepithelial Lesion; BK Polyomavirus
MeSH Terms: conditions — Salivary Gland Diseases | interventions — Ciprofloxacin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ciprofloxacin (Active Comparator): Active treatment twice daily for 28 days
  Interventions: Drug: Ciprofloxacin
- Placebo (Placebo Comparator): Placebo treatment twice daily for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin — Over encapsulated Ciprofloxacin 500 mg will be taken twice daily for 28 days.
  Other Names: Cipro
  Arms: Ciprofloxacin
Drug: Placebo — Placebo will over encapsulated to match active treatment, taken twice daily for 28 days.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to analyze BK viral infection in salivary gland diseases; specifically, to determine a definitive relationship between BK Virus and HIV associated salivary gland disease (HIVSGD). Participants are adults HIV+SGD+ who will be randomized 1:1 to receive BK Virus antiviral (ciprofloxacin) or placebo for 28 days. Salivary function/protein secretion will be correlated with BK polyomavirus titers. It is expected that patients with HIV+SGD+ will have elevated oral BK polyomavirus viral loads and will benefit from Ciprofloxacin.

DETAILED DESCRIPTION:
The study duration is 12 weeks with a baseline visit, a visit at 4 weeks and a visit at 12 weeks. At baseline participants are randomized to Ciprofloxacin or placebo and take the drug or placebo for 28 days. At subsequent visits BK polyomavirus presence and salivary gland function will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive with Salivary Gland Disease
* Ability to read and understand English

Exclusion Criteria:

* Allergy to the family of fluoroquinolones (including ciprofloxacin)
* Currently taking tizanidine
* Concurrently taking antiacids containing magnesium hydroxide or aluminum hydroxide
* Current use of Theophylline
* Previous tendon disorder such as Rheumatoid arthritis
* History of seizures
* Current use of phenytoin
* Current use of glyburide
* Current use of methotrexate
* Severe renal impairment (known creatinine clearance < 30 or on dialysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Webster-Cyriaque, DDS, PhD, Principal Investigator — The University of North Carolina School of Dentistry
Locations (1):
- The University of North Carolina School of Dentistry, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ciprofloxacin | Placebo
Started | 9 | 8
Completed | 8 | 7
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciprofloxacin | Placebo | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Full Range); unit: years] | 52.6 [37 to 69] | 52.3 [49 to 57] | 52.5 [37 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 3 | 1 | 4
  Black or African American | 5 | 4 | 9
  Asian | 0 | 1 | 1
  Hispanic or Latino | 0 | 2 | 2
  Other | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 8 | 17
BK Virus Status in Saliva [Count of Participants; unit: Participants] — Oral fluids will be assessed for evidence of BK Virus replication to determine whether Cipro administration inhibits BK Virus replication in participants with HIV associated salivary gland disease (HIVSGD). Oral fluids will be assessed by real-time polymerase chain reaction (PCR) to determine BK Virus status as positive or negative. Population: Data were not analyzed for one participant who discontinued
  Participants
    number analyzed (Participants) | 9 | 7 | 16
    BK Virus positive | 8 | 2 | 10
    BK Virus negative | 1 | 5 | 6
Unstimulated Salivary Flow Rate [Count of Participants; unit: Participants] — To determine salivary gland function at Baseline. After sitting at rest for 1 minute, participants collect drool using 50-mL conical tubes. The 5-minute unstimulated whole saliva flow rate recorded and collected. Salivary hypofunction is defined as unstimulated whole saliva flow rate ≤ 0.1 mL/min. Normal salivary function is defined as > 0.1 mL/min. Population: Data not collected because participant missed scheduled visit
  Participants
    number analyzed (Participants) | 9 | 7 | 16
    Normal salivary function | 4 | 1 | 5
    Salivary Hypofunction | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: BK Viral Status in Saliva at Week 4
Description: Oral fluids will be assessed for evidence of BK Virus replication to determine whether Cipro administration inhibits BK Virus replication in participants with HIVSGD. Oral fluids will be assessed by real-time PCR to determine BK Virus status as positive or negative.
Time Frame: Week 4
Population: Two participants withdrew prior to Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 8 | 7
Participants
  BK Virus positive | 3 | 6
  BK Virus negative | 5 | 1

2. Primary Outcome: BK Viral Status in Saliva at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: Two participants withdrew prior to Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 8 | 7
Participants
  BK Virus positive | 3 | 4
  BK Virus negative | 5 | 3

3. Secondary Outcome: Unstimulated Salivary Flow Rate at Week 4
Description: To determine whether salivary gland function is improved or restored with the administration of Cipro in participants with HIVSGD. After sitting at rest for 1 minute, participants collect drool using 50-mL conical tubes. The 5-minute unstimulated whole saliva flow rate recorded and collected. Salivary hypofunction is defined as unstimulated whole saliva flow rate ≤ 0.1 mL/min. Normal salivary function is defined as > 0.1 mL/min.
Time Frame: Week 4
Population: Two participants withdrew prior to Week 4 and one participant did not perform salivary flow collection.
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 8 | 6
Participants
  Normal salivary function | 3 | 1
  Salivary hypofunction | 5 | 5

4. Secondary Outcome: Unstimulated Salivary Flow Rate at Week 12
Description: To determine whether salivary gland function is improved or restored with the administration of Cipro in participants with HIVSGD. After sitting at rest for 1 minute, participants collect drool using 50-mL conical tubes. The 5-minute unstimulated whole saliva flow rate recorded and collected. Salivary hypofunction is defined as unstimulated whole saliva flow rate ≤0.1 mL/min. Normal salivary function is defined as >0.1 mL/min.
Time Frame: Week 12
Population: Two participants withdrew prior to Week 4 and two participants did not perform salivary flow collection.
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 7 | 6
Participants
  Normal salivary function | 3 | 1
  Salivary hypofunction | 4 | 5

5. Secondary Outcome: Number of Participants Reporting Dry Mouth "Yes/No" at Week 4
Description: Participants were asked "Have you noticed any change in your salivary glands or in the dryness of your mouth"
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 8 | 7
Participants
  Change = Yes | 2 | 1
  Change = No | 6 | 6

6. Secondary Outcome: Number of Participants Reporting Dry Mouth "Yes/No" at Week 12
Description: Participants were asked "Have you noticed any change in your salivary glands or in the dryness of your mouth"
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 8 | 7
Participants
  Change = Yes | 2 | 1
  Change = No | 6 | 6

ADVERSE EVENTS:
Arm/Group | Ciprofloxacin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 1/9 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciprofloxacin (N=9) | Placebo (N=8)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes